CLINICAL TRIAL: NCT05420038
Title: Do Bluetooth Noise Cancelling Headphones Improve the Quality of Care in Hearing Impaired Patients?
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0079
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Hearing Impairment
Keywords: hearing impairment; geriatric; headphones; noise-cancelling; hearing assistance; ophthalmic; refractive exams; ophthalmology; limited hearing; impaired hearing; quality of exam; Sound-Check hearing test
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Participants will be recruited by performing chart reviews of patients to be seen at University of Texas Medical Branch at Galveston Ophthalmology and Optometry Clinic. A sample size of at least 30 patients is needed (60 eyes). Patients aged 55 and higher will be further evaluated to meet the inclusion criteria. Patients meeting inclusion criteria will be provided with informed consent to participate in the study before their office visit. Patients will receive a consent briefing then asked to sign and date the informed consent form. Participants will then be randomized to undergo an eye exam and refractive exam with noise cancelling Bluetooth headphones for one eye and without for the other eye. Participants will fill out a written survey asking them to rate the quality of the eye exam with and without headphones.

Primary aim: Assess the quality improvement of Ophthalmic exam in geriatric patients with hearing loss with use of noise cancelling headphones with Bluetooth feature.

Secondary aims: 1)Compare the response to the standardized questions with and without Bluetooth noise cancelling headphones to determine their effectiveness in conducting Ophthalmic refractive exam.

2) Explore the ease of conducting refractive exam as reported by provider.

DETAILED DESCRIPTION:
Initial screening in this study will be conducted by performing chart reviews of the patients to be seen at University of Texas Medical Branch ophthalmology and optometry clinics between dates 05/09/2022 and 12/15/2022. Potential subjects will be provided with details about the study through debriefing about the informed consent before the start of their visit at University of Texas Medical Branch clinics. An option to participate in the study will be provided for recruitment by the principal investigator and the co-investigators. If potential subjects are not patients of the investigator or patients of the study team members, they will not be contacted by study staff unless they have been informed of the study by their medical provider and expressed an interest in receiving more information on the study or wish to enroll in the study. A sample size of at least 30 patients is needed (60 eyes). Patients aged 55 and higher will be further evaluated to meet the inclusion criteria. Patients meeting inclusion criteria will be provided with informed consent to participate in the study before their office visit. Patients will receive a consent briefing from the principal investigator or the co-investigators regarding the purpose of the study, number of people taking part in the study, procedures involved in the study, possible risks, potential benefits, reimbursement, alternative treatment, consent to leave study at any time, protection of patient information and privacy, and contact information for questions regarding the study. They will then be asked to sign and date the informed consent form. The signed consent forms will be stored in a locked file cabinet in room 3.420C of the University of Texas Medical Branch University Eye Clinic building. Patients who consent to participate in this study will then be randomized to undergo an eye exam and refractive exam with noise cancelling Bluetooth headphones for one eye and without for the other eye. The order in which the headphones are used will also be randomized by flipping a coin. Lastly, patients will fill out a written survey with a 3-point Likert scale with the following question:

How do you rate the quality of your eye exam today with headphones as compared to without headphones? 1) Better 2) No difference 3) Worse Primary aim: Assess the quality improvement of Ophthalmic exam in geriatric patients with hearing loss with use of noise cancelling headphones with Bluetooth feature.

Secondary aims: 1) Compare the response to the standardized questions with and without Bluetooth noise cancelling headphones to determine their effectiveness in conducting Ophthalmic refractive exam.

2) Explore the ease of conducting refractive exam as reported by provider.

ELIGIBILITY:
Inclusion Criteria:

* Participants are patients of University of Texas Medical Branch Ophthalmology and Optical clinics;
* patients of investigators;
* aged 55 years and above;
* participants with moderate hearing impairment or worse at baseline hearing grade of limited or impaired based on World Health Organization (WHO) hearing loss guidelines;
* participants with documented history of hearing loss;
* participants with no corrective procedures performed for hearing loss.

Exclusion Criteria:

* Participants with mild to no hearing impairment at baseline reported as hearing grade fair, good or excellent on the Sound-Check hearing test;
* participants with history of corrective procedure performed for hearing loss;
* participants with cognitive impairment;
* participants with visual impairment of best corrected visual acuity (BCVA) 20/100 or worse in either eye or patients with monocular vision;
* participants from vulnerable populations, such as prisoners.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Adults;
  * Elderly;
  * University of Texas Medical Branch Ophthalmology and Optical clinic patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Do Bluetooth Noise Cancelling Headphones Improve the Quality of Care in Hearing Impaired Patients? | 8 months
  Patients will fill out a written survey with a 3-point Likert scale with the following question: "How do you rate the quality of your eye exam today with headphones as compared to without headphone? 1) Better 2) No difference 3) Worse"

CONTACTS AND LOCATIONS:
Overall Officials: Praveena K Gupta, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chodosh J, Goldfeld K, Weinstein BE, Radcliffe K, Burlingame M, Dickson V, Grudzen C, Sherman S, Smilowitz J, Blustein J. The HEAR-VA Pilot Study: Hearing Assistance Provided to Older Adults in the Emergency Department. J Am Geriatr Soc. 2021 Apr;69(4):1071-1078. doi: 10.1111/jgs.17037. Epub 2021 Feb 11. PMID 33576037
- [Background] Sacco G, Gonfrier S, Teboul B, Gahide I, Prate F, Demory-Zory M, Turpin JM, Vuagnoux C, Genovese P, Schneider S, Guerin O, Guevara N. Clinical evaluation of an over-the-counter hearing aid (TEO First(R)) in elderly patients suffering of mild to moderate hearing loss. BMC Geriatr. 2016 Jul 9;16:136. doi: 10.1186/s12877-016-0304-4. PMID 27392722
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Bainbridge KE, Wallhagen MI. Hearing loss in an aging American population: extent, impact, and management. Annu Rev Public Health. 2014;35:139-52. doi: 10.1146/annurev-publhealth-032013-182510. PMID 24641557
- [Background] Nash SD, Cruickshanks KJ, Huang GH, Klein BE, Klein R, Nieto FJ, Tweed TS. Unmet hearing health care needs: the Beaver Dam offspring study. Am J Public Health. 2013 Jun;103(6):1134-9. doi: 10.2105/AJPH.2012.301031. Epub 2013 Apr 18. PMID 23597370
- [Background] Bentler R, Wu YH, Kettel J, Hurtig R. Digital noise reduction: outcomes from laboratory and field studies. Int J Audiol. 2008 Aug;47(8):447-60. doi: 10.1080/14992020802033091. PMID 18698521
- [Background] World Health Organization. Report of the informal working group on prevention of deafness and hearing impairment Programme planning, Geneva, 18-21 June 1991.
- [Derived] Glanzer BM, Ladki M, Chea MR, Hummel L, McKinnon B, Digbeu BDE, Merkley KH, Amin A, Gupta PK. Bluetooth Noise-Canceling Headphones Improve the Quality of Ophthalmic Exams in Patients With Hearing Loss: A Randomized Controlled Trial. Cureus. 2024 May 11;16(5):e60090. doi: 10.7759/cureus.60090. eCollection 2024 May. PMID 38860057